CLINICAL TRIAL: NCT04000009
Title: A 52-Week Open-Label Extension Study of Pimavanserin in Subjects With Major Depressive Disorder and Inadequate Response to Antidepressant Treatment
Brief Title: Extension Study of Pimavanserin in Subjects With Major Depressive Disorder and Inadequate Response to Antidepressant Treatment
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated for business reasons and not due to safety concerns.
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACP-103-055; 2018-003252-20 (EudraCT Number)
Record Dates: First submitted 2019-06-25; First posted 2019-06-27 (Actual); Results first posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Adjunctive Treatment of Major Depressive Disorder
MeSH Terms: interventions — pimavanserin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Drug - pimavanserin (Experimental): Pimavanserin 34 mg tablets
  Interventions: Drug: Pimavanserin

INTERVENTIONS:
Drug: Pimavanserin — Pimavanserin 34 mg (provided as 2×17 mg tablets) administered orally as a single dose once daily

SUMMARY:
To assess the safety and tolerability of long-term pimavanserin treatment in subjects with major depressive disorder and inadequate response to antidepressant treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Completed the antecedent study, Study ACP-103-054 or Study ACP-103-059
2. May benefit from longer term therapy with open-label pimavanserin treatment
3. If the subject is female, she must not be pregnant or breastfeeding. She must also be of nonchildbearing potential OR must agree to use acceptable methods of contraception

Exclusion Criteria:

1. Is determined to be inappropriate for the study
2. Has developed neurologic, cardiovascular, respiratory, gastrointestinal, renal, hepatic, hematologic, or other medical or mental disorder, including cancer or malignancies that would affect the patient's ability to participate in the program

Additional inclusion/exclusion criteria apply. Patients will be evaluated at screening to ensure that all criteria for study participation are met. Patients may be excluded from the study based on these assessments (and specifically, if it is determined that their baseline health and psychiatric condition do not meet all pre-specified entry criteria).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-02-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (71):
- United States (33):
  - CNS Network, Garden Grove, California
  - Behavioral Research Specialists, Glendale, California
  - Irvine Clinical Research, Irvine, California
  - Synergy San Diego, Lemon Grove, California
  - Pacific Research Partners, LLC, Oakland, California
  - NRC Research Institute, Orange, California
  - MCB Clinical Research centers, LLC, Colorado Springs, Colorado
  - Clinical Neuroscience Solutions ( CNS Healthcare)-Jacksonville, Jacksonville, Florida
  - Meridien Research, Maitland, Florida
  - Florida Research Center, Inc., Miami, Florida
  - CNS Health Care (Orlando), Orlando, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Synexus Clinical Research, Atlanta, Georgia
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Capstone Clinical Research, Libertyville, Illinois
  - Collective Medical Research, LLC, Prairie Village, Kansas
  - Adams Clinical, Watertown, Massachusetts
  - Integrative Clinical Trials, Brooklyn, New York
  - Social Psychiatry Research Institute (SPRI), Brooklyn, New York
  - Department of Psychiatry, Icahn School of Medicine at Mount Sinai, New York, New York
  - The Medical Research Network, LLC, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Charak Clinical Research Center, Garfield Heights, Ohio
  - Summit Research Network (Oregon) Inc., Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Clinical Neuroscience Solutions CNS Healthcare, Memphis, Tennessee
  - Research Strategies of Memphis, LLC, Memphis, Tennessee
  - Future Search Trials of Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Grayline Research Center, Wichita Falls, Texas
  - IPC Research, Waukesha, Wisconsin
- Finland (5):
  - ARTES Psykiatrinen Palvelukeskus Oy (Mederon Ltd.), Helsinki
  - Savon Psykiatripalvelu Oy, Kuopio
  - Oulu Mentalcare Oy, Oulu
  - Satakunnan Psykiatripalvelu Oy at Mehiläinen Pori, Pori
  - Psykiatri- ja psykologikeskus Mentoria, Tampere
- Poland (5):
  - Gabinet Lekarski Psychiatryczny Ireneusz Kaczorowski, Bełchatów
  - Przychodnia Śródmieście Sp. Z o.o., Bydgoszcz
  - Indywidualna Specijalistyczna Praktyka Lekarska Wiesław Jerzy Cubała, Gdansk
  - Nzop Mentis, Leszno
  - Zachodniopomorski Instytut Psychoterapii, Szczecin
- Russia (8):
  - Mental Health Research Center, Department #6, Moscow
  - St. Nicholas the Wonder Worker Psychiatric Hospital, Saint Petersburg
  - Psychoneurological Dispensary # 5, Saint Petersburg
  - City Narcology Hospital, Saint Petersburg
  - Samara Psychiatric Hospital, Samara
  - Saratov City Clinical Hospital #2 n.a. V.I. Razumovsky, Saratov
  - Regional Clinical Psychiatric Hospital of St. Sofia, Saratov
  - LION-MED, Voronezh
- Serbia (7):
  - Clinical Center of Serbia, Clinic for psychiatry, Belgrade
  - Clinical Hospital Center Dr Dragisa Misovic, Belgrade
  - Clinical Centre Nis, Clinic for Psychiatry, Gornja Toponica
  - Special hospital for psychiatric diseases "Kovin, Kovin
  - Clinical Center Kragujevac , Clinic for Psychiatry, Kragujevac
  - Clinical Center Kragujevac, Kragujevac
  - Centre for Mental Health Protecton, Clinical Center Nis, Niš
- Slovakia (3):
  - EPAMED s r.o., Košice
  - Liptovska nemocnice s poliklinikou MUDr. Ivana Stodolu, Psychiatricke oddelenie, Liptovský Mikuláš
  - Centrum Zdravia R.B.K., s.r.o., Svidník
- Flexivest Fourteen Research Centre, Unit 1, Durbanville Health Center, Durbanville, South Africa
- Ukraine (6):
  - Regional Centre of Psychosomatic Disorders based on Psychoneurology Department, Communal Institution Dnipropetrovsk Regional Clinical Hospital named after I.I. Mechnykov, Dnipro
  - Institute of neurology, Psychiatry and Narcology of NAMS of Ukraine, MC "Neuron", Kharkiv
  - Kyiv Railway Clinical Hospital № 1 of Branch "Health Center" of the Public joint stock company "Ukrainian Railway", Kyiv
  - Kherson Regional Psychiatric Hospital Department # 3 and # 10 Kherson region,, Stepanovka
  - Ternopil Regional Communal Clinical Psychoneurological Hospital, psychiatric department # 2 (men), psychiatric department # 6 (women), Ternopil State Medical University n.a. I.Y. Gorbachevskyy, Chair of Psychiatry, Narcology and Medical Psychology, Ternopil
  - Municipal Institution "Vinnytsya Regional Psychoneurological Hospital n.a. Acad. O.I.Yushchenko", Male Department #14, Female Department #15, Vinnytsya National Medical University n.a. M.I.Pyrogov, Department of Psychiatry, Narcology and Psychotherapeutic, Vinnytsia
- United Kingdom (3):
  - MAC Clinical Research- Blackpool, Blackpool
  - MAC Clinical Research Ltd.-Liverpool, Liverpool
  - MAC Clinical Research- Manchester, Manchester

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruited patients that had completed a previous study of pimavanserin, i.e. either study ACP-103-054 or ACP-103-059. It was planned to enroll about 420 patients in total.
  The study was terminated early by the Sponsor for business reasons due to the COVID-19 pandemic; there were no safety concerns contributing to study termination (see Caveats and Limitations). A total of 235 patients were enrolled and treated instead of the anticipated number of about 420 patients.
Pre-assignment Details: During the screening period, subjects were assessed for study eligibility and prohibited medications were discontinued when medically appropriate.
Groups:
- Pimavanserin: Pimavanserin 34 mg (administered as 2 x 17 mg pimavanserin tablets) once daily, for 52 weeks
Period: Overall Study
Arm/Group | Pimavanserin
Started | 235
Completed | 70
Not Completed | 165
Not completed — Adverse Event | 13
Not completed — Lack of Efficacy | 7
Not completed — Lost to Follow-up | 8
Not completed — Noncompliance with study drug | 4
Not completed — Physician Decision | 1
Not completed — Use of prohibited medication | 3
Not completed — Pregnancy | 1
Not completed — Withdrawal by Subject | 22
Not completed — Study terminated by sponsor | 98
Not completed — Not further specified | 8

BASELINE CHARACTERISTICS:
Population: All patients enrolled who received at least one dose of study medication
Arm/Group | Pimavanserin
Number analyzed (Participants) | 235
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (13.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 165
  Male | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 219
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 111
  Finland | 10
  Ukraine | 26
  Poland | 16
  South Africa | 1
  United Kingdom | 27
  Slovakia | 5
  Serbia | 13
  Russia | 26

OUTCOME MEASURES:

1. Primary Outcome: Treatment-emergent Adverse Events (TEAEs)
Description: Number of patients with treatment emergent AEs
Time Frame: 52 weeks
Population: All patients enrolled who received at least one dose of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | Pimavanserin
Number analyzed (Participants) | 235
Participants | 137

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | Pimavanserin
All-Cause Mortality (participants affected / at risk) | 0/235
Serious Adverse Events (participants affected / at risk) | 5/235
Other Adverse Events (participants affected / at risk) | 69/235
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pimavanserin (N=235)
Diverticular perforation (Gastrointestinal disorders) | 1 (1)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pimavanserin (N=235)
Diarrhoea (Gastrointestinal disorders) | 12 (13)
Nasopharyngitis (Infections and infestations) | 15 (17)
Urinary tract infection (Infections and infestations) | 12 (12)
Weight increased (Investigations) | 14 (14)
Headache (Nervous system disorders) | 29 (39)

LIMITATIONS AND CAVEATS:
This study was terminated early by the Sponsor for business reasons due to the COVID-19 pandemic; there were no safety concerns contributing to study termination. Patients were discontinued from the study and completed safety follow-up procedures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish the study results, relative to their own patients, only after review, comment and approval by the sponsor. No publication of confidential information shall be made without the sponsor's prior written consent. At least 60 days prior to submitting a manuscript or prior to any public presentation, a copy of the manuscript or presentation will be provided to the Sponsor for review and comment. The sponsor has 60 days to review and comment.

DOCUMENTS (2):
  • Study Protocol (2020-08-11): https://cdn.clinicaltrials.gov/large-docs/09/NCT04000009/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-11): https://cdn.clinicaltrials.gov/large-docs/09/NCT04000009/SAP_001.pdf